CLINICAL TRIAL: NCT04410068
Title: Comparison of Electric Heating Pad Versus Forced-air Warming to Prevent Inadvertent Perioperative Hypothermia: A Randomized Controlled Trial
Brief Title: Comparison of Electric Heating Pad Versus Forced-air Warming to Prevent Inadvertent Perioperative Hypothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-8860-I
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Temperature Change, Body; Hypothermia; Anesthesia
MeSH Terms: conditions — Body Temperature Changes; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electrical heating pad (Experimental): Electrical heating pad (WARMTAC device). Patients will be randomized to one arm.
  In this arm, the WARMTAC device will be conected and warmed to 41 degrees before patients lay down.
  Interventions: Device: WARMTAC
- forced-air warming device (Experimental): Forced-air warming device (3M device). In this arm, the 3M blanket will be conected to forced-air machine and warmed to 41 degrees before patients lay down.
  Interventions: Device: 3M Bair Hugger

INTERVENTIONS:
Device: WARMTAC — Randomization to one of the arms previous to surgery.
  Arms: Electrical heating pad
Device: 3M Bair Hugger — Randomization to one of the arms previous to surgery.
  Arms: forced-air warming device

SUMMARY:
Compare core body temperature after laparoscopic surgery using the forced air heating system versus the WARMTAC® (a carbon fiber electric blanket).

DETAILED DESCRIPTION:
In order to prevent perioperative hypothermia, we will compare two different heating sistems, one of them is an electric pad made with carbon fiber and the other system is a forced-air blanket. Both of them will be situated under the patient during all the laparoscopic surgey.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age at the time of the preoperative visit.
* Patients who will undergo elective laparoscopic surgery
* Patients who sign the informed consent indicating that they have been informed of all relevant aspects of the trial.

Exclusion Criteria:

* Axillary temperature> 37.5ºC
* Active infection
* Dysfunction of the autonomic system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Core body temperature | through study completion, an average of 12 months
  temperatured recorded in esophagus

SECONDARY OUTCOMES:
Rescues number | through study completion, an average of 12 months
  Compare number of rescues required by each system to avoid mild hypothermia
skin lesions | through study completion, an average of 12 months
  Detect possible skin complications related to heating

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Chanza, Physician, Principal Investigator — PSMar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calvo Vecino JM, Casans Frances R, Ripolles Melchor J, Marin Zaldivar C, Gomez Rios MA, Perez Ferrer A, Zaballos Bustingorri JM, Abad Gurumeta A; Grupo de trabajo de la GPC de Hipotermia Perioperatoria No Intencionada de la SEDAR. Clinical practice guideline. Unintentional perioperative hypothermia. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Dec;65(10):564-588. doi: 10.1016/j.redar.2018.07.006. Epub 2018 Nov 15. English, Spanish. PMID 30447894
- [Background] Matsuzaki Y, Matsukawa T, Ohki K, Yamamoto Y, Nakamura M, Oshibuchi T. Warming by resistive heating maintains perioperative normothermia as well as forced air heating. Br J Anaesth. 2003 May;90(5):689-91. doi: 10.1093/bja/aeg106. PMID 12697600
- [Background] Ng V, Lai A, Ho V. Comparison of forced-air warming and electric heating pad for maintenance of body temperature during total knee replacement. Anaesthesia. 2006 Nov;61(11):1100-4. doi: 10.1111/j.1365-2044.2006.04816.x. PMID 17042850
- [Background] John M, Crook D, Dasari K, Eljelani F, El-Haboby A, Harper CM. Comparison of resistive heating and forced-air warming to prevent inadvertent perioperative hypothermia. Br J Anaesth. 2016 Feb;116(2):249-54. doi: 10.1093/bja/aev412. PMID 26787794